CLINICAL TRIAL: NCT01418911
Title: Attachment Style of Type 2 Diabetics, and Cognitive, Social and Emotional Variables as Explanatory Factors of Adherence to Self-care Behavior and Diabetes Control
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assuta Hospital Systems (Other)
Responsible Party: Liza Cnaani, Maccabi Healthcare Services
Other Study IDs: 23/2011
Record Dates: First submitted 2011-08-16; First posted 2011-08-17 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2011-07

CONDITIONS: Type 2 Diabetes Patients
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- diabetes type 2: type 2 diabetes patients 40-70 years of age hebrew speaking members of maccabi healthcare services
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — questionnaire only

SUMMARY:
This study will expand the understanding of factors associated with adherence to self care and the diabetes control among diabetes type 2 patients. The theoretical framework of the study incorporates central variables from two theoretical models: a cognitive model of health behavior - "Health Belief Model", and the Stress and Coping model. The study is innovative in its focus on the association between the patient's attachment style and adherence to self care and diabetes control, a topic less studied among diabetes patients, in addition to cognitive, social and emotional variables. Further emphasis is upon a comparison of the study model between males and females.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* 40-70 years of age
* Hebrew speaking
* members of maccabi healthcare services

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: type 2 diabetes 40-70 years of age Hebrew speaking members of maccabi healthcare services
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Maccabi Healthcare Services, Tel Aviv, Israel, Israel